CLINICAL TRIAL: NCT00182169
Title: Randomized, Placebo Control, Clinical Trial Evaluating the Effect of Human Recombinant Growth Hormone in Patients With Severe Congestive Heart Failure. The Growth Hormone In Heart Failure Trial (GIFT)
Brief Title: Evaluation of the Effect of Human Recombinant Growth Hormone in Patients With Advanced Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004h00512
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2003-03

CONDITIONS: Heart Failure
Keywords: Severe heart failure; Growth hormone; exercise capacity; quality of life; cardiac function
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Drug: Human recombinant growth hormone

SUMMARY:
Prospective randomized, placebo controlled, clinical trial to evaluate the effect of human growth hormone supplementation compared with placebo to patients with severe heart failure for a duration of 6 months on exercise capacity, heart function and quality of life

ELIGIBILITY:
Inclusion Criteria:

Individuals with a diagnosis of CHF, NYHA functional class III or IV symptoms, an EF of < 35 % estimated on radionuclide angiography (RNA) or 2D echo within the last 6 months, and a 6 minute walk distance of less than 400 meters. Patients must be stabilized on "CHF" therapy at the time of randomization.

Exclusion Criteria:

1. Exercise limited by claudication, angina, neurological, pulmonary (FEV1 < 50%; FVC < 50%), or musculoskeletal disease.
2. Active known malignancy; remission of < 5 years from the diagnosis of malignancy; patients with recurrence of malignancy are to be withdrawn from the study.
3. Current diabetes with known retinopathy or patients with poorly controlled diabetes (ie. fasting glucose more than 13 mmol/l) or Type I diabetes mellitus.
4. Any other non-cardiac condition that substantially decreases survival.
5. Significant valvular stenosis or hypertrophic cardiomyopathy.
6. Unable to comply with GH injection.
7. Pregnancy or women of child bearing age not using adequate contraceptive means.
8. Unstable angina, acute myocardial infarct, cardiac surgery, or PTCA within 3 months.
9. Cor pulmonale.
10. Acute myocarditis.
11. Known need for cardiac surgery (e.g., valvular intervention, or CABG, or PTCA) within the next 6 months.
12. Clinical hypothyroidism or hyperthyroidism with biochemical corroboration (TSH > 7 or < 0.2) at screening.
13. Patients in need of urgent heart transplant within the next 6 months (patients on transplant list remain eligible).
14. Sustained ventricular tachycardia (lasting > 30 seconds) on screening Holter.
15. Significant liver disease (INR>1.4 off anticoagulant therapy; or AST, or ALT, or GGT, or alkaline phosphatase > 3X upper limit of normal; or bilirubin > 2X the upper limit of normal) at baseline.
16. Failure to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1997-07; Study Completion 2005-06

PRIMARY OUTCOMES:
6-minute walk test distance (functional capacity)measured at baseline, 3 months, and 6 months from the start of the study. Also measured at 3 months following discontinuation of therapy

SECONDARY OUTCOMES:
Cardiac Function measured with radionuclide angiography and echocardiography
Exercise capacity measured during treadmill testing (duration of exercise)
Quality of life measured with Minnesota Living with Heart Failure
Neurohormones
baseline, 3 months, and 6 months from the start of the study. Also measured at 3 months following discontinuation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Demers, MD, MSc, FRCPC, Study Director — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada